CLINICAL TRIAL: NCT03942627
Title: Promoting Maternal Mental Health and Wellbeing in Neonatal Intensive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB00159072; R34AT009615 (NIH)
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2020-10

CONDITIONS: Depressive Symptoms; Anxiety; Post-traumatic Stress Symptoms
Keywords: mindfulness; maternal depression
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Program (Experimental): The intervention consists of an introductory video in which a mindfulness expert explains the program's approach and models practices to increase women's comfort with the material, four audio-recorded mindfulness practices for mothers' use when the baby is in the NICU, each available in 5- and 10-minute versions, and a brief video and four additional audio mindfulness practices (each available in briefer and longer versions) for use by mothers during and following the transition home with the baby.
  Interventions: Behavioral: Mindfulness Program
- Infant Health Education Program (Placebo Comparator): The intervention consists of an introductory video explaining the program's approach, four audio recordings providing education about infant health and development, each available in 5- and 10-minute versions, and a brief video and four additional educational recordings (each available in briefer and longer versions) for use by mothers during and following the transition home with the baby.
  Interventions: Behavioral: Infant Health Education Program

INTERVENTIONS:
Behavioral: Mindfulness Program — The intervention consists of two brief videos (one introducing the NICU portion of the program and one introducing the portion of the program addressing the transition home), as well as a series of mindfulness practices delivered via audio recordings to assist mothers in managing stress during the NICU stay and another series for the transition home.
  Arms: Mindfulness Program
Behavioral: Infant Health Education Program — The active control condition consists of two brief videos (one introducing the NICU portion of the program and one introducing the portion of the program addressing the transition home), as well as a series of audio recordings providing information on infant health and development for mothers to use during the NICU stay and another series for the transition home.
  Arms: Infant Health Education Program

SUMMARY:
This small randomized pilot study will evaluate feasibility and preliminary outcomes of an audio-delivered mindfulness program to reduce psychological distress for mothers with an infant in neonatal intensive care, as compared with an active control condition.

DETAILED DESCRIPTION:
An estimated 400,000-480,000 infants in the U.S. with serious medical conditions are cared for in neonatal intensive care units (NICUs) each year. Maternal stress exposure related to infants' NICU stays is an under-appreciated public health problem with negative implications for maternal and child health and wellbeing. Flexible, effective intervention strategies have potential to improve maternal mental health and parenting, promoting positive emotional and behavioral outcomes for both mothers and infants.

In the investigators' successful pilot research, the investigators developed an audio-delivered mindfulness program to help NICU mothers reduce rumination and worry, cultivate a state of calm awareness, and promote self care. In this small randomized pilot study, the investigators will randomly assign mothers with an infant in the neonatal intensive care unit (NICU) to receive either the mindfulness intervention or an active control program (audio-delivered education on infant care and development).

This study will evaluate feasibility of all key research aspects, including recruitment, randomization, intervention and control conditions, and assessments, in preparation for a future larger-scale study. This study will also assess preliminary intervention outcomes to identify potential program benefits.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18 to 50 years old
* mother of an infant currently being treated in the Johns Hopkins Hospital or Johns Hopkins Bayview Medical Center NICU
* able to speak English

Exclusion Criteria:

* known to have serious psychopathology
* infant medically unstable/ progress is poor

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms as assessed by the Patient Health Questionnaire (PHQ)-8 | 2 weeks
  Self-reported depressive symptoms over the last 2 weeks. Each of the 8 items is scored 0 (not at all) to 3 (nearly every day), yielding a total between 0 and 24. Higher scores mean more depressive symptoms.
Anxiety symptoms as assessed by the Generalized Anxiety Disorder - 7 (GAD-7) | 2 weeks
  Self-reported anxiety symptoms over the last 2 weeks. Each of the 7 items is rated from 0 (not at all) to 3 (nearly every day), yielding a total between 0 and 21. Higher scores mean more anxiety.

SECONDARY OUTCOMES:
Trauma symptoms as assessed by the Stanford Acute Stress Reaction Questionnaire (SASRQ) | 2 weeks
  31-item self-report measure of trauma symptoms. Items 1-30 are rated from 0 (not experienced) to 5 (very often experienced). Item 31 asks how many days symptoms were experienced since giving birth, ranging from no days to 5 or more days. Higher scores mean more frequent experience of trauma symptoms.
Perceived stress as assessed by the Perceived Stress Scale - NICU (PSS-NICU) | Up to 2 weeks
  Self-report measure of perceived stress related to the NICU containing 4 sub scales, each with items rated on a scale of 1 (not at all stressful) to 5 (very stressful). Higher scores mean more stress.
Sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | 4 weeks
  Self-reported measure assessing sleep quality
Coping as assessed by the Brief Cope Scale | Up to 2 weeks
  28-item self-reported measure of coping strategies. Items are rated on a scale ranging from 1 ("I usually don't do this at all") to 4 ("I usually do this a lot")

CONTACTS AND LOCATIONS:
Overall Officials: Erica Sibinga, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mendelson T, McAfee C, Damian AJ, Brar A, Donohue P, Sibinga E. A mindfulness intervention to reduce maternal distress in neonatal intensive care: a mixed methods pilot study. Arch Womens Ment Health. 2018 Dec;21(6):791-799. doi: 10.1007/s00737-018-0862-x. Epub 2018 Jun 5. PMID 29872924